CLINICAL TRIAL: NCT04850924
Title: Alex Storm: Acute Stress Manifestations' Description in French Pediatric Population
Brief Title: Emergency Psychological Intervention With Children: Alex Storm
Acronym: ALEX
Status: Completed | Type: Observational
Sponsor: Fondation Lenval (Other)
Responsible Party: Sponsor
Other Study IDs: 21-HPNCL-01
Record Dates: First submitted 2021-04-12; First posted 2021-04-20 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Psychological Trauma
MeSH Terms: conditions — Psychological Trauma

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- children impact by the Alex storm
  Interventions: Other: evaluation psychological trauma

INTERVENTIONS:
Other: evaluation psychological trauma — 9 classes of symptoms to be evaluated

SUMMARY:
Alex storm hits France, especially the French Riviera, from September 30, 2020 to October 3, 2020. A lot of people have been impacted by this event. Among these people, 116 children have been taking care by the medico-psychological emergency unit and have been assessed by child psychiatrists or by psychologists.

DETAILED DESCRIPTION:
Alex storm hits France from September 30, 2020 to October 3, 2020. On October 2, several valley in the Nice hinterland were devastated by this natural disaster. Nine people died during this storm and hundreds of families were affected (house washed away or uninhabitable). This led to emergency evacuations on October 3 of several families. The inhabitants of some villages have been subjected to prolonged stress (lack of water and electricity, difficulty in supplying food, fear of another storm). These villages were isolated for a period varying from fifteen days to over three months. These people are particularly exposed to psychological consequences.

Between October 3 and October 30, the CUMP (medico-psychological emergency unit) was mobilized to provide psychological first aid to these families. Among those seen in emergency 116 children were taken care of. In order to assess the immediate symptoms of the children, the investigators used an assessment sheet specific to the developmental ages of the children.

All children seen in an emergency between October 3 and October 30, 2020 were assessed by child psychiatrists or by psychologists trained in emergency and pediatric psychological trauma.

ELIGIBILITY:
Inclusion Criteria:

* children impacted by the Alex storm
* children seen in an emergency between October 3 and October 30, 2020
* children were assessed by child psychiatrists or by psychologists trained in emergency and pediatric psychological trauma

Exclusion Criteria:

* children whose parents refused to the processing of their data

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children aged between 0 to 18 years. Impacted by the Alex Storm and evacuated to Nice airport
Sampling Method: Non-Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2021-01-18 (Actual); Primary Completion 2021-02-26 (Actual); Study Completion 2021-02-26 (Actual)

PRIMARY OUTCOMES:
measure of risk developing post-traumatic stress disorder | at inclusion
  A questionnaire assessing symptoms in the acute phase. 9 classes of symptoms to be evaluated..
  Anxiety - Sadness / Cries - Mutism / Apartness - Passiveness - Agitation / Panic / Disorganization - Somatization - Developmental regression / Excessive attachment to caregiver - Verbalization of fear - Sleep disorders All symptoms are assessed by scoring presence (1) or absence (0). The total score is calculated out of 9 and refers to the risk of later developing post-traumatic stress disorder (PTSD) (0 = very low risk; 9 = very high risk)

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpitaux Pédiatriques de Nice CHU-Lenval, Nice, France

REFERENCES:
- [Derived] Richez A, Gindt M, Battista M, Nachon O, Menard ML, Askenazy F, Fernandez A, Thummler S. Storm Alex: acute stress responses in the pediatric population. Eur J Psychotraumatol. 2022 May 11;13(1):2067297. doi: 10.1080/20008198.2022.2067297. eCollection 2022. PMID 35599977